CLINICAL TRIAL: NCT02498834
Title: Using Question Prompt Lists During Pediatric Asthma Visits to Increase Adolescent Involvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-2628; CDR-1402-09777 (Other: PCORI)
Record Dates: First submitted 2015-06-24; First posted 2015-07-15 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: Asthma
Keywords: Communication; provider; caregiver; adolescent
MeSH Terms: conditions — Asthma; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Video and Question Prompt List (Experimental): Parents and adolescents in this group will watch a short educational video in English or Spanish on an iPad about the importance of encouraging adolescents to ask questions and to be involved during their pediatric asthma visits to improve their self-management skills. Also, the adolescents in this group will be handed a question prompt list to complete, which will be collected after the medical visit.
  Interventions: Behavioral: Educational Video and Question Prompt List
- Control group (No Intervention): Standard of care will be used

INTERVENTIONS:
Behavioral: Educational Video and Question Prompt List — Educational Video and Question Prompt List
  Arms: Educational Video and Question Prompt List

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial with English and Spanish-speaking adolescents to compare the effectiveness of an adolescent "asthma question prompt list" with a supportive educational video intervention with usual care.

The hypothesis of this study is that by showing the parents and adolescents the educational video and then providing the adolescents with the one-page "asthma question prompt lists" to use during their visits will improve: (a) asthma control, (b) adolescent self-efficacy in managing asthma, and (c) adolescent quality-of-life.

DETAILED DESCRIPTION:
The study uses a randomized controlled trial design stratified by provider to assess the impact of an adolescent "asthma question prompt list" combined with a supportive educational video emphasizing the importance of adolescent involvement and question-asking on communication during pediatric visits. This application is based on Social Cognitive Theory. Self-confidence or self-efficacy is a central component of Social Cognitive Theory (SCT) Application of Social Cognitive Theory (SCT) in asthma populations has shown that technical advice from providers is one external factor that can improve asthma management self-efficacy. Additionally, personal beliefs, such as outcome expectations, and family factors, such as parent and adolescent responsibility for asthma self-management, have been shown to affect adolescent self-efficacy and disease management outcomes. Prior work has found that adolescent self-efficacy in asthma management correlates strongly with health status, adherence, asthma medication device technique, asthma symptoms, and impact of illness on the family.

All adolescents will have their medical visits audio recorded. The adolescent will be interviewed after his/her medical visit while his/her caregiver/parent completes a survey at the time of study enrollment. This same procedure will be used when the adolescent and caregiver/parents return for the 6- and 12-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* ages 11 to 17 years;
* speak and read English or Spanish;
* have persistent asthma;
* are present for an acute or follow-up asthma visit or a well-child visit;
* and have previously visited the clinic at least once for asthma.

Adolescents' parents will be eligible if they are at least 18 years of age, speak and read English or Spanish, and are the legal guardian of the adolescent.

Exclusion Criteria:

* present for gastrointestinal complaints or other non-asthma related acute illness.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 359 (Actual)
Dates: Start 2015-07; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betsy L Sleath, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolin at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Educational Video and Question Prompt List | Control Group
Started | 185 | 174
Completed | 175 | 164
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Video and Question Prompt List | Control Group | Total
Number analyzed (Participants) | 185 | 174 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (1.9) | 13.2 (1.9) | 13.2 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 78 | 154
  Male | 109 | 96 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 19 | 45
  Not Hispanic or Latino | 159 | 155 | 314
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 17 | 41
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 71 | 63 | 134
  White | 60 | 70 | 130
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 30 | 20 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 185 | 174 | 359
Number of Participants Achieving Asthma Control [Count of Participants; unit: Participants] — This will be measured via the 5-item Asthma Control Test, responses are summed to indicate a score ranging from 5 (poor asthma control) to 25 (complete asthma control). A higher score means a better outcome. A score of above 19 is considered "well-controlled".
  Participants
    Controlled | 101 | 105 | 206
    Not controlled | 84 | 69 | 153
Adolescent asthma management self-efficacy score [Mean (Standard Deviation); unit: score on a scale] — Adolescent asthma management self-efficacy was measured using a 14-item scale that has been shown to have a reliability of 0.87. Prior work in asthma has found asthma management self-efficacy to change in response to an intervention. Scores range from 14 to 70 and a higher score means a better outcome.
  score on a scale | 55.9 (8.0) | 56.0 (8.2) | 55.9 (8.1)
Asthma quality-of-life score [Mean (Standard Deviation); unit: score on a scale] — Adolescent quality-of-life was measured as a continuous variable. The investigators used the standardized version of the Juniper pediatric asthma quality-of-life questionnaire. The questionnaire contains 23 items and has a reliability of 0.84. Scores can range from 1.0 to 7.0, and a higher score means a better outcome.
  score on a scale | 5.7 (1.2) | 5.8 (1.2) | 5.7 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Asthma Control
Description: This will be measured via the 5-item Asthma Control Test, responses are summed to indicate a score ranging from 5 (poor asthma control) to 25 (complete asthma control). A higher score means a better outcome. A score of above 19 is considered "well controlled".
Time Frame: 12 month follow-up
Population: One intervention group patient was excluded because they had to leave immediately after the final visit and did not complete the 12-month survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Video and Question Prompt List | Control Group
Number analyzed (Participants) | 174 | 164
Participants
  Controlled | 121 | 128
  Not controlled | 53 | 36

2. Primary Outcome: Adolescent Asthma Management Self-efficacy Score
Description: Adolescent asthma management self-efficacy was measured using a 14-item scale that has been shown to have a reliability of 0.87. Prior work in asthma has found asthma management self-efficacy to change in response to an intervention. Scores range from 14 to 70 and a higher score means a better outcome.
Time Frame: 12 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Educational Video and Question Prompt List | Control Group
Number analyzed (Participants) | 174 | 164
score on a scale | 58.9 (8.6) | 59.7 (7.2)

3. Primary Outcome: Asthma Quality-of-life Score
Description: Adolescent quality-of-life was measured as a continuous variable. The investigators used the standardized version of the Juniper pediatric asthma quality-of-life questionnaire. The questionnaire contains 23 items and has a reliability of 0.84. Scores can range from 1.0 to 7.0, and a higher score means a better outcome.
Time Frame: 12 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Educational Video and Question Prompt List | Control Group
Number analyzed (Participants) | 174 | 164
score on a scale | 6.1 (1.2) | 6.2 (0.98)

ADVERSE EVENTS:
Time Frame: Up to approximately 1 year following enrollment
Arm/Group | Educational Video and Question Prompt List | Control Group
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/174
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/174
Other Adverse Events (participants affected / at risk) | 0/185 | 0/174

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT02498834/Prot_SAP_000.pdf